CLINICAL TRIAL: NCT03654846
Title: Video-assisted Telephone CPR With the EmergencyEye-Software - a Pilot Study - Proof of Concept
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, PD Dr. med. Wolfgang A. Wetsch, PI, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EmergencyEye-POC
Record Dates: First submitted 2018-08-25; First posted 2018-08-31 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Test of EmergencyEye functionality in real environment, comparison with conventional emergency call.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional emergency call (No Intervention): Emergency call with conventinal cell phone:
  * verbal description of location
  * telephone-assisted CPR
- EmergencyEye emergency call (Experimental): Emergency call with EmergencyEye App on cell phone:
  * automated geolocalisation
  * video-assisted CPR
  Interventions: Device: EmergencyEye

INTERVENTIONS:
Device: EmergencyEye — EmergencyEye Smartphone App
  Arms: EmergencyEye emergency call

SUMMARY:
Technical advance as broad-bandwidth wireless internet coverage and the ubiquity utilization of smartphones has opened up new possibilities which surpass the normal audio-only telephony. High quality and real-time video-telephony is now feasible. However until now this technology hasn't been deployed in the emergency respond service.

In the hope of helping the detection of the cardiac arrest, offer the possibility to evaluate and correct via a video-instructed CPR (V-CPR) and to facilitate a fast localization of the emergency site, a new software (EmergencyEye®/RAMSES®) was developed which enables the dispatcher a video-telephony with the callers mobile terminal (smartphone) if suitable.

This technology hasn't been tested in a randomized controlled trial in real environment conditions yet. This is to be done in this study.

DETAILED DESCRIPTION:
Technical advance as broad-bandwidth wireless internet coverage and the ubiquity utilization of smartphones has opened up new possibilities which surpass the normal audio-only telephony. High quality and real-time video-telephony is now feasible. However until now this technology hasn't been deployed in the emergency respond service.

In the hope of helping the detection of the cardiac arrest, offer the possibility to evaluate and correct via a video-instructed CPR (V-CPR) and to facilitate a fast localization of the emergency site, a new software (EmergencyEye®/RAMSES®) was developed which enables the dispatcher a video-telephony with the callers mobile terminal (smartphone) if suitable, and automated localisation of the caller.

This technology hasn't been tested in a randomized controlled trial in real environment conditions yet. This is to be done in this study.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* cardiovascular diseases
* pulmonary diseases
* pregnancy
* all other conditions that make CPR impossible

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-08-25 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Recognition of CPR quality through video transmission | 1 minute of CPR
  Recognition of CPR quality (3 conditions are randomized in each CPR, i.e. Frequency, Compression Depth, Compression Point) in Video-assisted CPR

SECONDARY OUTCOMES:
Time to first chest compression | Study duration (approx. 1 minute)
  Time measured from the beginning of the emergency call to the first chest compression
Precision of Geolocalisation | Study duration (approx. 1 minute)
  Precision of Geolocalisation, i.e. difference between verbally localized and automatically localized (aGPS) respondes to emergency call. Difference in runtimes of dispatched ambulances will be calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Critical Care Medicine, University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided